CLINICAL TRIAL: NCT02572401
Title: Reducing the Risk of HIV/STD Infection Among African American Men
Brief Title: Steering Together in a New Direction: Reducing the Risk of HIV/STD Among African American Men
Acronym: STAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 810971; R01MD004075 (NIH)
Record Dates: First submitted 2015-09-28; First posted 2015-10-08 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Human Immunodeficiency Virus (HIV); Sexually Transmitted Disease (STD)
Keywords: Human immunodeficiency virus; Sexually transmitted disease; Behavioral intervention; Randomized controlled trial; Text messages; Social cognitive theory; Theory of planned behavior; Sexual behavior; African Americans; Men
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Sexual Behavior; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- HIV Risk Reduction Only (Experimental): STAND HIV Risk Reduction Intervention. Participants will not receive the Text Messaging Intervention.
  Interventions: Behavioral: STAND HIV Risk Reduction Intervention
- No-Intervention No-Text Message Control (No Intervention): Participants do not receive the STAND HIV Risk Reduction Intervention or the Text Messaging Intervention.
- HIV Risk Reduction and Text Messaging (Experimental): STAND HIV Risk Reduction Intervention and Text Messaging Intervention. Participants will receive the intervention and text messages.
  Interventions: Behavioral: STAND HIV Risk Reduction Intervention; Behavioral: Text Messaging Intervention
- Text Messaging Only (Experimental): Text Messaging Intervention. Participants will receive the text messages but not the STAND HIV Risk Reduction Intervention.
  Interventions: Behavioral: Text Messaging Intervention

INTERVENTIONS:
Behavioral: STAND HIV Risk Reduction Intervention — STAND HIV Risk Reduction Intervention, designed to increase consistent condom use and reduce other sexual risk behaviors, is implemented in small groups over 2 weekly 135-minute sessions. It draws on social cognitive theory, the reasoned action approach, and focus groups, a prospective survey, and an intervention pilot test with African American men. It contains culturally appropriate video clips, interactive activities, brainstorming, role-playing, and discussions designed to affect hypothesized mediators of risk-reducing behavior, including outcome expectancies about the effects of condom use on sexual enjoyment; self-efficacy and skill to have condoms available and to stop to use condoms or refuse unsafe sex even when aroused; and self-efficacy and skill to negotiate condom use.
  Other Names: HIV Risk Reduction Intervention
  Arms: HIV Risk Reduction Only; HIV Risk Reduction and Text Messaging
Behavioral: Text Messaging Intervention — Text Messaging Intervention participants receive text messages designed to increase the consistent use of condoms and to reduce other sexual risk behaviors. They receive 3 times a week text messages that ask about their sexual behavior and condom use that day and are asked to respond with either a 1 or 2 numeric response to indicate yes or no. Based on their responses, they receive either an affirming, pro safe-sex text message or a cautionary text against unprotected sex.
  Arms: HIV Risk Reduction and Text Messaging; Text Messaging Only

SUMMARY:
African American men have by far the highest rates of HIV in the US, but there are few randomized controlled trials (RCTs) of interventions to dissuade heterosexually active African American men from engaging sexual risk behavior. This research seeks to address this gap in the behavioral intervention literature. That self-initiated behavior change, as well as intervention-induced behavior change, is often short-lived, eroding over time, is widely known; accordingly, this research also seeks to test a strategy to sustain intervention efficacy. In a RCT, African American men 18 to 45 years reporting recent unprotected intercourse with a woman will be randomized to the Steering Together in a New Direction (STAND) HIV Risk Reduction Intervention or a No-Intervention Control Condition. To test a strategy to sustain intervention effects, the men also will be randomized to receive or not receive individually tailored text messages. The theoretical basis of the interventions is social cognitive theory and the reasoned action approach, which is an extension of the theory of planned behavior and the theory of reasoned action. Men will complete self-report measures via audio computer-assisted self-interviewing at baseline and immediately post and 6 and 12 months post-intervention. The trial will test whether the STAND HIV Risk Reduction Intervention as compared with the No-Intervention Control Condition, increases consistent condom use, the primary outcome. Secondary outcomes include unprotected intercourse, multiple sexual partners, insertive anal intercourse, and proportion condom-protected intercourse. The trial will also test whether STAND's efficacy is greater among men in the Text Messaging Intervention compared with men not receiving text messages. This will provide information on the utility of a low-cost strategy to extend an intervention's efficacy. Finally, the study will test for mediation of intervention effects: the hypothesis that STAND affects outcome expectancies and self-efficacy, which, in turn, affect consistent condom use.

DETAILED DESCRIPTION:
HIV/AIDS has had a devastating impact on African Americans, who have the highest rates of HIV/AIDS as compared with Whites, Hispanics, Asians, and Native Americans. Although African Americans comprise only 13% of the US population, more than 40% of people living with HIV/AIDS in the US are African American-some 192,277 people. New diagnoses of HIV/AIDS underscore the epidemic's impact on African Americans. Almost 50% of the people newly diagnosed with HIV/AIDS in the 33 states with confidential name-based HIV infection reporting in 2006 were African Americans. The overall rate of newly diagnosed cases was 19 cases per 100,000, but among African Americans, it was 68 per 100,000. The estimated rates of HIV/AIDS in 2006 were higher among African American men (121 per 100,000) as compared with White men (17 per 100,000), Latino/Hispanic men (51 per 100,000), and African American women (57 per 100,000). Heterosexual exposure is a key HIV transmission category among African Americans. To be sure, the largest number of estimated cases of HIV/AIDS among African American men fell in the men who have sex with men (MSM) HIV-transmission category. However, the second largest number of cases was attributed to heterosexual transmission, with the injection-drug-use HIV-transmission category ranking third. Moreover, heterosexual exposure was a more important HIV-transmission category among African American men than among other men. It accounted for 23% of HIV/AIDS cases among African American men, but 19% among Hispanic men and only 7% of cases among White men. Furthermore, among African American women, who comprised over 60% of the women with HIV/AIDS in 2006, heterosexual exposure was by far the most important transmission category, accounting for 83% of cases. Heterosexual exposure is especially important in Philadelphia, Pennsylvania, where the proposed study will be conducted. According to the Philadelphia Department of Public Health, among African American men, heterosexual exposure surpassed male-to-male contact as the modal exposure category in 2006, 2007, and 2008.

Furthermore, another important health disparity affecting African Americans particularly in urban areas is the high rate of sexually transmitted disease (STD). About 47% of the cases of Chlamydia trachomatis (CT) reported to Centers for Disease Control and Prevention (CDC) in 2006 occurred in African Americans. The CT rate was 7 times higher among African American women than among White women. The Neisseria gonorrhea rate was 25 times higher among African American men than among White men and 14 times higher among African American women than among their White counterparts. Despite the high rate of heterosexual exposure to HIV and the high rates of other STDs in African American men and women, little research has focused on interventions targeting heterosexually active men.

Sexual Risk Behavior among Heterosexually Active African American Men

Two key behaviors that increase risk of STD, including HIV, are failing to use condom consistently and having multiple sexual partners. Although unmarried African American men were more likely to report consistent condom use than were their Hispanic or White counterparts, which may reflect recognition of higher risk of STD among African American men, a large percentage of African American men (47%) risked exposure to HIV and other STDs. Moreover, consistent condom use declined substantially with increasing age, from 68% in those 15 to 19 years of age, to 31% in those 25 to 29 years of age, and to only 26% in those 40 to 44 years of age. In the National Survey of Family Growth, among men 15-44 years of age, unmarried African American men were more likely to have had 4 or more partners in the past year (13%) compared with White (6%) and Hispanic men (7%).

Interventions to Reduce Risk of Heterosexual Transmission of HIV in African American Men

Whether one considers the domestic or international literature, few randomized controlled trials (RCTs) of interventions have focused on risk of heterosexual transmission of HIV among men. Of particular concern is the paucity of trials on the efficacy of risk-reduction interventions specifically targeting African American men. A systematic review of HIV/STD risk-reduction interventions found that only 12 of 1157 intervention studies worldwide were conducted on males only, and only 4 focused exclusively on African American adult men. A more recent review of interventions to reduce heterosexual transmission of HIV among African Americans identified 38 RCTs, but only 7 targeted males only and 2 of the 7 focused on adolescent boys. Thus, only 5 of the 38 trials focused specifically on African American men. Combining the studies identified in these 2 reviews yields only 6 trials specifically on heterosexual transmission among African American adult men and only 1 focused on the general population of heterosexual men. A recent clinic-based study on 266 African American men 18 to 29 years of age diagnosed with an STD is more encouraging. At 3-month follow-up, those randomized to a single session one-on-one intervention reported fewer unprotected sex acts than did those who received standard clinical care. In addition, medical-records review revealed that the intervention participants were less likely to acquire a new STD by 6 months post-intervention than were the control men. Although the few existing studies are an important first step in beginning to develop interventions for African American men, there is still an important gap in the literature as noted by Seal and Ehrhardt who asserted that heterosexual men's sexual and reproductive health is often exclusively viewed in the context of their female partners. They called for interventions that focus on men's health and consider men's heterosexual behavior as a starting point in intervention development.

Sustaining Intervention-Induced Behavior Change

As evidence accumulates for the benefits of behavioral interventions it is also clear that often the effects are short lived. The present study will test the efficacy of a relatively inexpensive strategy to sustain behavior change. Many strategies have been employed. The inclusion of booster sessions in intervention programs has been suggested as a strategy to extend their effects, a strategy consistent with relapse prevention approaches that have been employed in substance-abuse reduction and smoking cessation programs. Several HIV risk-reduction intervention studies have incorporated boosters in their interventions, but the existing studies do not provide clear evidence for the efficacy of boosters per se, because they were not designed to compare the effects of an HIV/STD risk-reduction intervention with a booster to the effects of that same intervention without the booster. In addition to booster sessions, there may be other effective methods for extending intervention effects. Telephone counseling programs have been shown to help smokers who are in the process of quitting. Periodic mailings have also been found to be more effective than a telephone hot line in preventing relapse among former cigarette smokers.

This study will test whether text messages extend an HIV risk-reduction intervention's efficacy. The use of text messaging has several advantages. It is relatively inexpensive, possibly even more cost effective than other phone or print-based interventions. Participants do not have to return for another intervention session, facilitators do not have to conduct the sessions, and no space must be made available. Text messages are delivered almost immediately and can be stored in the recipient's phone, accessible at a time that suits him. Tailored messages are more efficacious than are messages that are not tailored, and text messages can be individually tailored to promote condom use to men who fail to use them for different reasons. Pew surveys reveal that a great majority of African Americans own cell phones, African Americans are more intense and frequent users of all the phones' capabilities than are Whites, and more African Americans than Whites use text messaging. Although RCTs of text-messaging interventions have reported significant effects on healthful behaviors, including reduced cigarette smoking, increased adherence to insulin regimens in diabetics, and increased medical appointment keeping, no trials have examined whether text messaging can enhance the efficacy of an HIV risk-reduction intervention.

The study will utilize a RCT design. Participants will be recruited through advertising in a local free newspaper, through community based organizations that serve African Americans, through recruitment flyers at universities, bars, health clubs, and health fairs, and through face-to-face recruitment at social and sports events and activities expecting a high turnout of African American men. Computer-generated random number sequences will be used to randomize them to the Steering Together in a New Direction (STAND) HIV Risk Reduction Intervention or a No-Intervention Control Condition and to receive or not receive a Text Messaging Intervention. Participants will complete assessments via audio computer-assisted self-interviewing before the intervention and immediately post and 6 and 12 months post-intervention administered by data collectors blind to the participants randomly assigned condition. The trial will test whether the STAND intervention increases the consistent use of condoms and decreases other sexual risk behaviors compared with the no-intervention control group, whether the text messages are efficacious, and whether the efficacy of the STAND intervention is enhanced among men who receive the text messages.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 45 years
* Self-identify as African American or Black
* Born a male
* Report having intercourse with a woman in the past 60 days without using a condom

Exclusion Criteria:

* Report having intercourse with only 1 female partner in the past 60 days and being in a committed relationship with her for 6 or more months
* Plan to relocate beyond a reasonable distance from the study in the next 18 months or do not have an address where he can receive mail
* Report participating in an intervention research study on how to reduce HIV risks or negotiate safer sex in the previous 12 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 391 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B Jemmott III, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV Risk Reduction Only: STAND HIV Risk Reduction Intervention. Participants will not receive the Text Messaging Intervention.
  STAND HIV Risk Reduction Intervention: STAND HIV Risk Reduction Intervention, designed to increase consistent condom use and reduce other sexual risk behaviors, is implemented in small groups over 2 weekly 135-min sessions. It draws on social cognitive theory, the reasoned action approach, and focus groups, a prospective survey, and an intervention pilot test with African American men. It contains culturally appropriate video clips, interactive activities, brainstorming, role-playing, and discussions designed to affect hypothesized mediators of risk-reducing behavior, including outcome expectancies about the effects of condom use on sexual enjoyment; self-efficacy and skill to have condoms available and to stop to use condoms or refuse unsafe sex even when aroused; and self-efficacy and skill to negotiate condom use.
- HIV Risk Reduction and Text Messaging: STAND HIV Risk Reduction Intervention and Text Messaging Intervention. Participants will receive the intervention and text messages.
  STAND HIV Risk Reduction Intervention: STAND HIV Risk Reduction Intervention, designed to increase consistent condom use and reduce other sexual risk behaviors, is implemented in small groups over 2 weekly 135-min sessions. It draws on social cognitive theory, the reasoned action approach, and focus groups, a prospective survey, and an intervention pilot test with African American men. It contains culturally appropriate video clips, interactive activities, brainstorming, role-playing, and discussions designed to affect hypothesized mediators of risk-reducing behavior, including outcome expectancies about the effects of condom use on sexual enjoyment; self-efficacy and skill to have condoms available and to stop to use condoms or refuse unsafe sex even when aroused; and self-efficacy and skill to negotiate condom use.
  Text Messaging Intervention:
Period: Overall Study
Arm/Group | HIV Risk Reduction Only | No-Intervention No-Text Message Control | HIV Risk Reduction and Text Messaging | Text Messaging Only
Started | 97 | 98 | 98 | 98
Completed | 92 | 90 | 89 | 88
Not Completed | 5 | 8 | 9 | 10
Not completed — Lost to Follow-up | 5 | 8 | 9 | 9
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Risk Reduction Only | No-Intervention No-Text Message Control | HIV Risk Reduction and Text Messaging | Text Messaging Only | Total
Number analyzed (Participants) | 97 | 98 | 98 | 98 | 391
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 97 | 98 | 98 | 98 | 391
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.18 (8.28) | 27.65 (8.63) | 27.73 (8.28) | 28.42 (8.60) | 27.75 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 97 | 98 | 98 | 98 | 391
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 4 | 2 | 11
  Not Hispanic or Latino | 95 | 95 | 94 | 96 | 380
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 95 | 94 | 94 | 95 | 378
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 2 | 3 | 2 | 1 | 8
  Unknown or Not Reported | 0 | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 97 | 98 | 98 | 98 | 391

OUTCOME MEASURES:

1. Primary Outcome: Consistent (100%) Condom Use
Description: A binary variable reflecting whether or not the participant reports using a condom every time he had vaginal or anal intercourse with a woman in the previous 3 months. It will be based on a comparison of the number of protected intercourse acts and the number of intercourse acts. Men who report at least one intercourse act and whose number of reported protected acts equals their number of acts use condoms during 100% of intercourse acts and will be defined as practicing consistent condom use. Men who report at least one intercourse act and whose reported number of protected acts is less than their number of acts will be coded as not practicing consistent condom use. Separate binary variables reflect consistent condom use with steady partners and casual partners analyzed as a repeated outcome.
Time Frame: Baseline, 6 months, 12 months post-intervention
Population: Participants providing primary outcome data at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Risk Reduction Only | No-Intervention No-Text Message Control | HIV Risk Reduction and Text Messaging | Text Messaging Only
Number analyzed (Participants) | 67 | 56 | 74 | 71
Participants
  Baseline steady partners: number analyzed (Participants) | 48 | 35 | 53 | 52
  Baseline steady partners | 9 | 6 | 7 | 7
  6 mo steady partners: number analyzed (Participants) | 44 | 35 | 50 | 52
  6 mo steady partners | 6 | 5 | 8 | 9
  12 mo steady partners: number analyzed (Participants) | 40 | 37 | 53 | 43
  12 mo steady partners | 10 | 5 | 12 | 11
  Baseline casual partners: number analyzed (Participants) | 50 | 43 | 59 | 49
  Baseline casual partners | 26 | 12 | 27 | 15
  6 mo casual partners: number analyzed (Participants) | 36 | 34 | 40 | 36
  6 mo casual partners | 13 | 12 | 13 | 17
  12 mo casual partners: number analyzed (Participants) | 30 | 28 | 41 | 31
  12 mo casual partners | 11 | 13 | 16 | 12
Statistical Analysis 1: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; The primary analysis tested the efficacy of the HIV risk reduction intervention by comparing the HIV Risk Reduction Only and HIV Risk Reduction and Text Messaging Arms to the Text Messaging Only and No-Intervention No Text Message Control Arms. This is a test of the main effect of the HIV risk reduction intervention; Test type: Superiority; p < .05, Poisson regression; Adjusted for baseline of the criterion and time of follow-up assessment (6 vs. 12 months); Risk Ratio (RR) = 0.84, 95% CI 2-sided [.59 to 1.21] — The numerator is the treatment
Statistical Analysis 2: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; This analysis tested the efficacy of the text messaging intervention by comparing the HIV Risk Reduction and Text Messaging and Text Messaging Only Arms to the HIV Risk Reduction Only and No-Intervention No Text Message Control Arms. This is a test of the text messaging main effect; Test type: Superiority; p < .05, Poisson regression; Adjusted for baseline of the criterion and time of follow-up assessment (6 vs. 12 months); Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.69 to 1.42] — The numerator is the treatment
Statistical Analysis 3: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; The analysis tested whether text messaging enhanced the effects of the HIV risk reduction intervention by comparing the HIV Risk Reduction and Text Messaging and No-Intervention No Text Message Arms to the Text Messaging Only and HIV Risk Reduction Only Arms. This is a test of the interaction between the two types of interventions; Test type: Superiority; p < .05, Poisson regression; Adjusted for baseline of the criterion, time of follow-up assessment (6 vs. 12 months), and the HIV x Time and Text Messaging x Time interactions; Risk Ratio (RR) = .72, 95% CI 2-sided [.35 to 1.49] — The numerator is the treatment

2. Secondary Outcome: Unprotected Intercourse
Description: A binary variable indicating whether the participants reported having intercourse in the past 90 days without using a condom. It was constructed by subtracting the sum of the condom-protected intercourse acts from the total number of intercourse acts in the past 90 days. If the difference was one or greater the participant was coded as having unprotected intercourse; if the difference was zero or if the person reported no intercourse in the past 90 days, the person was coded as not having unprotected intercourse. Calculated separately for steady partners and casual partners and analyzed as a repeated outcome.
Time Frame: Baseline, 6 months, 12 months post-intervention
Population: Participants providing the outcome measure at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Risk Reduction Only | No-Intervention No-Text Message Control | HIV Risk Reduction and Text Messaging | Text Messaging Only
Number analyzed (Participants) | 90 | 89 | 89 | 87
Participants
  Baseline steady partners: number analyzed (Participants) | 90 | 88 | 89 | 87
  Baseline steady partners | 42 | 31 | 48 | 47
  6 mo steady partners: number analyzed (Participants) | 85 | 85 | 85 | 81
  6 mo steady partners | 46 | 39 | 45 | 46
  12 mo steady partners: number analyzed (Participants) | 82 | 85 | 84 | 83
  12 mo steady partners | 38 | 42 | 43 | 35
  Baseline casual partners: number analyzed (Participants) | 59 | 59 | 66 | 54
  Baseline casual partners | 31 | 41 | 37 | 37
  6 mo casual partners: number analyzed (Participants) | 85 | 85 | 85 | 81
  6 mo casual partners | 23 | 26 | 28 | 22
  12 mo casual partners: number analyzed (Participants) | 82 | 85 | 84 | 83
  12 mo casual partners | 22 | 17 | 25 | 21
Statistical Analysis 1: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .05, Poisson regression; Adjusted for baseline of the criterion and time of follow-up assessment (6 vs. 12 months); Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.92 to 1.18] — The numerator is the treatment
Statistical Analysis 2: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < .05, Poisson regression; Adjusted for baseline of the criterion; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.90 to 1.16] — The numerator is the treatment
Statistical Analysis 3: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < .05, Poisson regression; [statistical method as in outcome 1, analysis 3]; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.86 to 1.42] — The numerator is the treatment

3. Secondary Outcome: Multiple Partners
Description: Participants whose number of intercourse partners in the past 90 days was 2 or greater are coded as having multiple partners, and those who reported having 0 or 1 intercourse partners in the past 90 days are coded as not having multiple partners.
Time Frame: Baseline, 6 months, 12 months post-intervention
Population: Participants who provide data on the outcome measure at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Risk Reduction Only | No-Intervention No-Text Message Control | HIV Risk Reduction and Text Messaging | Text Messaging Only
Number analyzed (Participants) | 92 | 89 | 89 | 87
Participants
  Baseline | 61 | 52 | 59 | 61
  6 mo: number analyzed (Participants) | 86 | 85 | 85 | 81
  6 mo | 40 | 39 | 43 | 45
  12 mo: number analyzed (Participants) | 84 | 85 | 84 | 83
  12 mo | 40 | 33 | 46 | 36
Statistical Analysis 1: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .05, Poisson regression; Adjusted for baseline of the criterion; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.89 to 1.24] — The numerator is the treatment
Statistical Analysis 2: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs Text Messaging Only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < .05, Poisson regression; Adjusted for baseline of the criterion and time of follow-up assessment (6 vs. 12 months); Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.94 to 1.30]; The numerator is the treatment
Statistical Analysis 3: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < .05, Poisson regression; [statistical method as in outcome 1, analysis 3]; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.76 to 1.47] — The numerator is the treatment

4. Secondary Outcome: Insertive Anal Intercourse
Description: A binary variable indicating whether the participant reported having insertive anal intercourse in the past 90 days. Measured separately for steady partners and casual partners and analyzed as a repeated outcome.
Time Frame: Baseline, 6 months, 12 months post-intervention
Population: Participants who provided data on the outcome measure at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Risk Reduction Only | No-Intervention No-Text Message Control | HIV Risk Reduction and Text Messaging | Text Messaging Only
Number analyzed (Participants) | 92 | 90 | 89 | 88
Participants
  Baseline steady partners | 9 | 7 | 11 | 8
  6 mo steady partners: number analyzed (Participants) | 86 | 86 | 85 | 82
  6 mo steady partners | 10 | 7 | 8 | 10
  12 mo steady partners: number analyzed (Participants) | 84 | 86 | 84 | 84
  12 mo steady partners | 11 | 12 | 8 | 10
  Baseline casual partners | 12 | 13 | 11 | 7
  6 mo casual partners: number analyzed (Participants) | 86 | 86 | 85 | 82
  6 mo casual partners | 7 | 6 | 6 | 4
  12 mo casual partners: number analyzed (Participants) | 84 | 86 | 84 | 84
  12 mo casual partners | 3 | 5 | 5 | 3
Statistical Analysis 1: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .05, Poisson regression; Adjusted for baseline of the criterion and time of follow-up assessment (6 vs. 12 months); Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.73 to 1.48] — The numerator is the treatment
Statistical Analysis 2: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < .05, Poisson regression; Adjusted for baseline of the criterion and time of follow-up assessment (6 vs. 12 months); Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.71 to 1.45] — The numerator is the treatment
Statistical Analysis 3: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < .05, Poisson regression; [statistical method as in outcome 1, analysis 3]; Risk Ratio (RR) = 1.02, 95% CI 2-sided [.50 to 2.08] — The numerator is the treatment

5. Secondary Outcome: Proportion Condom-protected Intercourse
Description: The denominator is the number intercourse acts in the past 90 days and the numerator is the number of condom-protected intercourse acts in the past 90 days. Calculated separately for steady partners and casual partners and analyzed as a repeated outcome.
Time Frame: Baseline, 6 months, 12 months post-intervention
Population: Participants who provided data on the outcome measure at baseline and at least one post-intervention assessment.
Measure: Mean (Standard Deviation); unit: proportion
Arm/Group | HIV Risk Reduction Only | No-Intervention No-Text Message Control | HIV Risk Reduction and Text Messaging | Text Messaging Only
Number analyzed (Participants) | 67 | 56 | 74 | 71
proportion
  Baseline steady partners: number analyzed (Participants) | 48 | 35 | 53 | 52
  Baseline steady partners | .51 (.38) | .40 (.42) | .34 (.40) | .42 (.41)
  6 mo steady partners: number analyzed (Participants) | 44 | 35 | 50 | 52
  6 mo steady partners | .39 (.42) | .43 (.40) | .45 (.42) | .45 (.43)
  12 mo steady partners: number analyzed (Participants) | 40 | 37 | 53 | 43
  12 mo steady partners | .46 (.42) | .39 (.40) | .41 (.44) | .44 (.45)
  Baseline casual partners: number analyzed (Participants) | 50 | 43 | 59 | 49
  Baseline casual partners | .71 (.38) | .60 (.37) | .66 (.41) | .59 (.39)
  6 mo casual partners: number analyzed (Participants) | 36 | 34 | 40 | 36
  6 mo casual partners | .56 (.44) | .58 (.40) | .64 (.42) | .64 (.45)
  12 mo casual partners: number analyzed (Participants) | 30 | 28 | 41 | 31
  12 mo casual partners | .69 (.37) | .64 (.42) | .64 (.40) | .58 (.43)
Statistical Analysis 1: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .05, Regression, Linear; Adjusted for baseline of the criterion and time of follow-up assessment (6 vs. 12 months); Mean Difference (Final Values) = .001, 95% CI 2-sided [-0.078 to 0.080]
Statistical Analysis 2: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs Text Messaging Only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < .05, Regression, Linear; Adjusted for baseline of the criterion and time of follow-up assessment (6 vs. 12 months); Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.082 to 0.076]
Statistical Analysis 3: Comparison: HIV Risk Reduction Only vs No-Intervention No-Text Message Control vs HIV Risk Reduction and Text Messaging vs Text Messaging Only; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < .05, Regression, Linear; [statistical method as in outcome 1, analysis 3]; Mean Difference (Final Values) = -0.009, 95% CI 2-sided [-0.167 to 0.149]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | HIV Risk Reduction Only | No-Intervention No-Text Message Control | HIV Risk Reduction and Text Messaging | Text Messaging Only
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/98 | 0/98 | 1/98
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/98 | 0/98 | 0/98
Other Adverse Events (participants affected / at risk) | 0/97 | 0/98 | 0/98 | 0/98

LIMITATIONS AND CAVEATS:
The outcome measures are self-reported; hence, they may be biased by socially desirable responding or problems of memory. The participants were not randomly selected; hence the findings may not generalize to the target population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes